CLINICAL TRIAL: NCT04344457
Title: An Open-Label, Single-Arm, Phase II Study to Evaluate the Efficacy and Safety of Oral Hydroxychloroquine, Indomethacin and Zithromax in Subjects Positive With SARS-CoV-2 With Mild Symptoms
Brief Title: Evaluate the Efficacy and Safety of Oral Hydroxychloroquine, Indomethacin and Zithromax in Subjects With Mild Symptoms of COVID-19
Acronym: COVID-19
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Perseverance Research Center, LLC (Other)
Collaborators: Athena Medical Group (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIZ-PRC-COVID-19
Record Dates: First submitted 2020-04-08; First posted 2020-04-14 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; Indomethacin; Azithromycin

STUDY DESIGN:
Intervention Model Description: Open label, single arm study
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Hydroxychloroquine — 200 mg PO BID 7 days
Drug: Indomethacin — 50 mg PO TID 14 Days
Drug: Zithromax Oral Product — 500 mg PO QD 3 Days

SUMMARY:
Currently there are no US Food and Drug Administration (FDA)-approved drugs specifically for the treatment of patients with COVID-19. At present, clinical management includes infection prevention and control measures, as well as supportive care, including supplementary oxygen and mechanical ventilatory support when indicated. An array of drugs approved for other indications as well as several investigational drugs are being studied in several hundred clinical trials that are underway across the globe; however, currently there are no clinical trials available to patients in Arizona.

This study will determine if a specific drug cocktail can improve clinical outcomes in patients with confirmed Mild SARS-CoV-2

DETAILED DESCRIPTION:
COVID-19 has become a massive threat to public health worldwide. Current estimates suggest that the novel coronavirus (SARS-CoV-2) is both highly contagious (estimated reproductive rate, 2-3) and five to fifty-fold more lethal than seasonal influenza (estimated mortality rate, 0.5-5%); therefore, interventions to decrease the incidence and severity of COVID-19 are emergently needed. In Maricopa County there has yet to be a clinical trial to evaluate people who are SARS-CoV-2 positive with mild symptoms. This study will measure the improvement of COVID-19 disease status as measured by time (days) required from initiation of treatment to improvement of clinical status from mild to symptom free on 14 days of a cocktail therapy of Hydroxychloroquine, Indomethacin and Zithromax.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years of age
2. Willing and able to provide written informed consent prior to performing study procedures
3. Confirmed Sars-CoV2 infection by PCR
4. Have mild symptoms of Sars-CoV2
5. Must show documentation of Sars-CoV2 to screening visit
6. Must have had recent hematology and chemistry results
7. Must be able to take heart rate daily
8. Must agree to Skype/Facetime daily
9. Must agree to take temperature daily
10. Must agree not to enroll in another study of an investigational agent prior to completion of Day 14 of treatment.

Exclusion Criteria:

1. Known to be allergic to research drugs or drug excipients
2. Incapable of providing informed consent
3. Participation in any other clinical trial of an experimental treatment for Sars-CoV2 infection
4. Pregnancy, possible pregnancy or breast feeding
5. Prolonged QT interval (>450)
6. Moderate to severe symptoms of Sars-CoV2
7. Renal failure
8. Hepatic failure
9. NSAID use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-04-16 (Actual); Primary Completion 2020-06-20 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Improvement of clinical status | up to 28 days
  measured by time (days) required from initiation of treatment to improvement of clinical status from mild to symptom free

SECONDARY OUTCOMES:
Time of clinical recovery of fever | up to 15 days
  the time of normalization of fever as measured by daily temperature ( - ≤36.6°C or -axilla, ≤37.2 °C oral or ≤37.8°C rectal or tympanic)
Time of clinical recovery of cough | up to 28 days
  the time of alleviation of cough as measured by self reported visual analog scale (VAS) cough scale. 1=no cough, 2-3=cough sometimes, 4-6=have a cough but can still do things, 7-8=persistent cough, prevents from doing things, 9-10=cough presents a great deal of discomfort
Safety as determined by changes in QTC intervals measured by ECG | up to 15 days
  to determine the safety of these therapies in combination
Safety as determined by presence of side effects | up to 15 days
  to assess the presence or absence of side effects and whether they are tolerable
Time to improvement | up to 28 days
  improvement in Wisconsin Upper Respiratory Symptom Survey (WURSS-44) 0 to 7 scale, with 0 = Do not have, 1 = Very mild, 3 = Mild, 5 = Moderate, 7 = Severe

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Gaither, NP, Principal Investigator — Athena Medical Group; Nicole C. Hank, PhD, MCR, MHSM, Study Director — Perseverance Research Center
Locations (2):
- United States (2):
  - Perseverance Research Center, Scottsdale, Arizona
  - Covidcraz 19, Llc, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.prcresearchaz.com